CLINICAL TRIAL: NCT05114538
Title: Improving the Part C Early Intervention Service Delivery System for Children with ASD: a Randomized Clinical Trial
Brief Title: Improving the Part C Early Intervention Service Delivery System for Children with ASD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Michigan State University (Other); Rush University Medical Center (Other); University of Massachusetts, Boston (Other)
Responsible Party: Principal Investigator, Wendy Stone, Professor, Psychology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00009835; 1R01MH122727-01 (NIH)
Record Dates: First submitted 2021-10-06; First posted 2021-11-10 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Enrollment: 440 parent-child dyads; 160 providers (anticipated)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RIT Training Group (Experimental): Providers in the RIT group (n=80) will receive intensive training (online tutorial, 2-day workshop, and virtual coaching and feedback in the field) in RIT and parent coaching and will be required to achieve fidelity prior to enrolling families from their caseload. They will then be asked to use the intervention with enrolled families for a minimum of 3 months. One intervention session per month for each enrolled family will be videotaped and scored for fidelity. Providers will receive monthly consultation from RIT trainers while these families are in the active treatment phase.
  Interventions: Behavioral: Reciprocal Imitation Training
- Treatment as Usual (No Intervention): Providers in the TAU group (n=80) will have three sessions videotaped and scored for each enrolled family to assess treatment differentiation. To incentivize agency participation, RIT training will be provided to the TAU group and other providers when data collection is complete.

INTERVENTIONS:
Behavioral: Reciprocal Imitation Training — RIT is a relatively straightforward, brief NDBI. It employs four simple strategies to target motor imitation and IJA during play: (1) contingent imitation of the child's verbal and nonverbal behavior, (2) linguistic mapping, (3) direct elicitation of object and gesture imitation following the child's interest, and (4) contingent reinforcement. It has been used at low intensities (e.g., 1-3 hours per week) over short periods of time (e.g., 10-12 weeks) to produce robust changes in pivotal skills. It is easy to learn and can be implemented with fidelity by undergraduate-level therapists with limited backgrounds in ASD, as well as by parents and siblings.
  Arms: RIT Training Group

SUMMARY:
Despite strong consensus that early, specialized intervention for children with autism spectrum disorder (ASD) can have a dramatic impact on outcomes, the public health system's capacity to provide such services is severely challenged by the rapid rise in ASD prevalence. The goal of this research project is to increase timely and equitable access to ASD-specialized early intervention during the critical first three years of life by capitalizing on the existing infrastructure of the Part C Early Intervention (EI) system, which is publicly funded and available in all states in the United States. This project will train EI providers to use an evidence-based, parent-mediated intervention that can improve child and family outcomes as well as mitigate the long-term substantial economic costs associated with ASD.

DETAILED DESCRIPTION:
The long-term goal of this study is to improve services and outcomes for children with early social communication challenges and/or ASD by increasing the capacity to provide appropriately specialized treatment within an existing infrastructure: the Part C Early Intervention (EI) service delivery system. Part C is publicly funded, available throughout the United States, and serves children under age 3 who have developmental delays or disabilities. Currently, the effectiveness of EI services is limited by high practice variation and infrequent use of evidence-based interventions. We are conducting a randomized controlled trial (RCT) to examine the effectiveness of training EI providers to deliver Caregiver-Implemented Reciprocal Imitation Teaching (CI-RIT) to children showing early social communication challenges. RIT is a naturalistic developmental behavioral intervention (NDBI) that is ideally suited for EI settings because it is low intensity, play-based, easy to learn and implement, and can be taught to families for their independent use (in the form of CI-RIT), thus increasing intervention dosage.

This RCT will employ a hybrid type 1 effectiveness/ implementation design and will use a unique mixed methods approach to gather evidence that will be essential for implementing RIT at scale, pending positive trial results. The sample includes a target of 20 EI agencies (across 4 U.S. States), 160 EI providers and 440 families of children with early social communication challenges, which not only provides a robust sample size, but also affords the opportunity to assess the generalizability of this approach across regions that vary in their implementation of Part C services. EI providers will be randomly assigned to the RIT training group (n=80) or treatment as usual (TAU; n=80). Providers in both groups will identify 2-5 children in their caseload who are 16-33 months old with early social communication delays (target n=220 children per group). Intensive, state-of-the art, multimethod assessment technology will be used to measure the impact of the intervention. Child and family assessments will be conducted at baseline, 4 months after enrollment, and 9 months after enrollment. Importantly, this study will examine putative mechanisms through which RIT improves clinically-relevant outcomes. In sum, this study will generate the evidence necessary to implement RIT at scale, thereby increasing the capacity of the existing EI system to deliver effective, evidence-based intervention to the rapidly growing population of children who show early social communication challenges.

The objectives of the RISE study are as follows:

1. To test the effectiveness of CI-RIT as delivered by community-based EI providers for improving child- and caregiver/family-level outcomes. We hypothesize that compared to TAU, children working with CI-RIT providers will demonstrate greater improvements in motor imitation and joint attention at T2 (4-months post-baseline), and language and social communication at T3 (9-months post-baseline). We also hypothesize that compared to TAU, caregivers working with CI-RIT providers will show greater improvements in contingent responsivity, RIT strategy use, parenting efficacy, and family quality of life.
2. To analyze the mechanisms by which CI-RIT improves outcomes. We hypothesize that changes in children's social communication and language outcomes will be serially mediated by gains in: (a) caregiver contingent responsivity and caregiver RIT strategy use, and (b) children's motor imitation and joint attention. We hypothesize that changes in caregiver/family outcomes will be mediated by gains in caregiver contingent responsivity, caregiver RIT strategy use, child motor imitation, and child joint attention.
3. To prepare for implementation at scale by identifying potential sources of practice variation to inform refinement of RIT training and development of quality assurance protocols. Triangulating evidence from video observations of EI sessions, EI provider self-reports, and qualitative interviews, we will use the Model for Adaptation Design (MADI) framework (32) to characterize the modifications to RIT that providers make (MADI domain 1), to identify potential mediating or moderating factors of these modifications (e.g., relationship to fidelity, rationale) (MADI domain 2), and to explore whether all or certain modifications influence implementation outcomes (e.g., ongoing fidelity, treatment acceptability) (MADI domain 3). This robust implementation evaluation will provide relevant information for improving the delivery of all NDBIs in the Part C system.

ELIGIBILITY:
Inclusion Criteria:

* Child has a diagnosis of ASD or displays early social communication challenges
* Child receives ≥ 1 weekly session with the participating provider (not co-treated with another provider)
* Caregiver is present during EI sessions
* Caregiver is the biological parent or custodial guardian
* Caregiver is at least 18 years of age
* Caregiver speaks either English or Spanish

Exclusion Criteria

- the child has visual, hearing, or motor conditions that would compromise his/her ability to participate in RIT or assessments

Ages: 16 Months to 33 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 440 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Weighted Frequency of Intentional Communication | Change from baseline to 9 months
  The Weighted Frequency of Intentional Communication coding protocol will be used to measure expressive communication during a virtual administration of an adapted version of the Communication Play Protocol (CPP; Adamson et al., 2004).
Vineland-3 | Change from baseline to 9 months
  The Communication and Social Domain standard scores from the Vineland-3 will be used to measure child social communication
Parenting Efficacy Scale (PES) | Change from baseline to 9 months
  The PES Total Score will be used to measure parenting efficacy.
Initiation of Joint Attention | Change from baseline to 4 months
  An adapted version of the ESCS coding protocol (Roos et al., 2008) will be used to measure initiation of joint attention within a virtual administration of an adapted version of the Communication Play Protocol (CPP; Adamson et al., 2004).
Unstructured Imitation | Change from baseline to 4 months
  An adapted version of the UIA coding protocol (Ingersoll, 2012) will be used to measure spontaneous motor imitation within a virtual administration of an adapted version of the Communication Play Protocol (CPP; Adamson et al., 2004).
Adapted Motor Imitation Scale (MIS) | Change from baseline to 4 months
  Elicited motor imitation will be assessed using a virtually-administered version of the Motor Imitation Scale (MIS).
The Parenting Interactions with Children: Checklist of Observations Linked to Outcomes (PICCOLO) | Change from baseline to 4 months
  The PICOOLO coding protocol will be used to measure caregiver responsivity from caregiver- child interaction videos.
CI-RIT Caregiver Fidelity Form | Change from baseline to 4 months
  The CI-RIT Caregiver Fidelity Form will be used to measure caregiver fidelity of the RIT strategies from caregiver- child interaction videos.

SECONDARY OUTCOMES:
MacArthur Bates Communicative Development Inventory (MCDI) | Change from baseline to 9 months
  The total number of words said on the MCDI will be used to measure expressive vocabulary.
Language Environment Analysis (LENA) Vocal Complexity | Change from baseline to 9 months
  Child vocal complexity will be based on recorded language using LENA Software.
Language Environment Analysis (LENA) Vocal Contingency | Change from baseline to 9 months
  Child reciprocal vocal contingency will be based on recorded language using the LENA software.
Parent Interview for Autism-Clinical Version (PIA-CV) | Change from baseline to 9 months
  Social Communication domains from the PIA-CV will be used to measure child social communication.
Family Life Impairment Scale (FLIS) | Change from baseline to 9 months
  The FLIS Total Impairment Score will be used to measure family well-being.

OTHER OUTCOMES:
Parenting Stress Index-Short Form | Baseline
  Parenting stress will be measured using the Parenting Stress Index-Short Form (PSI-SF) [Moderator]
Developmental Play Assessment (DPA | Baseline
  Total number of differentiated acts on toys will be assessed using a virtually-administered version of the Developmental Play Assessment (DPA) [Moderator]
Vineland-3 | Baseline
  The Adaptive Behavior Composite score will be used to measure child developmental level [Moderator]

CONTACTS AND LOCATIONS:
Overall Officials: Wendy L Stone, PhD, Principal Investigator — University of Washington
Locations (4):
- United States (4):
  - Rush University Medical Center, Chicago, Illinois
  - University of Massachusetts Boston, Boston, Massachusetts
  - Michigan State University, East Lansing, Michigan
  - Carol A Schubert, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nadwodny N, Yoder PJ, Ingersoll BR, Wainer AL, Stone WL, Eisenhower A, Carter AS; RISE Research Network. The Language ENvironment Analysis (LENA) System in Toddlers With Early Indicators of Autism: Test-Retest Reliability and Convergent Validity With Clinical Language Assessments. Autism Res. 2025 Aug;18(8):1568-1579. doi: 10.1002/aur.70062. Epub 2025 Jun 2. PMID 40452405
- [Derived] Wainer AL, Edmunds SR, Carter AS, Stone WL, Sheldrick RC, Broder-Fingert S, Stern YS, Harrington E, V Ibanez L, Ingersoll B. A hybrid type I randomized effectiveness-implementation trial of a Naturalistic Developmental Behavioral Intervention in the Part C early intervention system: study protocol. BMC Pediatr. 2025 Apr 1;25(1):263. doi: 10.1186/s12887-025-05587-8. PMID 40170032
- [Derived] Ingersoll B, Howard M, Oosting D, Carter AS, Stone WL, Berger N, Wainer AL, Britsch ER; RISE Research Network. Adapting measures of motor imitation for use by caregivers in virtual contexts: Reliability, validity, and sensitivity to change. Autism Res. 2025 Jan;18(1):122-132. doi: 10.1002/aur.3267. Epub 2024 Nov 21. PMID 39569704
- [Derived] Ingersoll B, Espinel A, Nauman J, Broder-Fingert S, Carter AS, Sheldrick RC, Stone WL, Wainer AL. Using virtual multiteam systems to conduct a multisite randomized clinical trial in the part C early intervention system: Benefits, challenges, and lessons learned. Contemp Clin Trials. 2024 Aug;143:107585. doi: 10.1016/j.cct.2024.107585. Epub 2024 May 29. PMID 38821261